CLINICAL TRIAL: NCT05031689
Title: Green Banana Peel Extract for Melasma Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, Adriana Rodrigues dos Anjos Mendonça, Principal Investigator, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Melasma
Record Dates: First submitted 2021-08-20; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Melasma
Keywords: Melasma; banana; skin; sunscreen
MeSH Terms: conditions — Melanosis | interventions — Drug Compounding

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPF 30 and Placebo (Placebo Comparator): Control Group will use SPF 30 sunscreen plus pharmaceutical formulation without green banana peel extract
  Interventions: Biological: SPF 30 sunscreen plus pharmaceutical formulation without green banana peel extract
- SPF 30 and pharmaceutical formulation with green banana peel (Active Comparator): In Study Group, in addition to the SPF 30 sunscreen, a pharmaceutical formulation containing the extract of the green banana peel will be used.
  Interventions: Biological: SPF 30 sunscreen and pharmaceutical formulation containing green banana peel extract

INTERVENTIONS:
Biological: SPF 30 sunscreen plus pharmaceutical formulation without green banana peel extract — Control Group will use SPF 30 sunscreen plus pharmaceutical formulation without green banana peel extract
  Arms: SPF 30 and Placebo
Biological: SPF 30 sunscreen and pharmaceutical formulation containing green banana peel extract — Study Group In addition to the SPF 30 sunscreen, a pharmaceutical formulation containing green banana peel extract will be used.
  Arms: SPF 30 and pharmaceutical formulation with green banana peel

SUMMARY:
To develop and evaluate a pharmaceutical formula based on green banana peel extract for the treatment of melasma.

DETAILED DESCRIPTION:
Objective: to develop and evaluate a pharmaceutical formula based on green banana peel extract for the treatment of melasma. Methods: it will be a clinical, interventional, longitudinal study, random sampling, Sample will have 60 patients divided into two groups. In the Control Group, SPF 30 sunscreen plus pharmaceutical formulation without green banana peel extract will be used, and in the Study Group, in addition to SPF 30 sunscreen, pharmaceutical formulation containing green banana peel extract will be used. Patients will undergo treatment for 90 days, evaluated every 30 days through clinical evaluation and MELASQol.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with melasma.
* Patients aged 18 years or over and 60 years or less.
* Patients who agree to participate in the study. -

Exclusion Criteria:

* Patients who have other types of facial hyperchromia.
* Patients who give up, for any reason, to continue treatment.
* Patients who have any type of allergic reaction to the product.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Clinical analysis of Melasma | 3 months
  Analysis of the skin affected by Melasma will be performed with Melasma Area Severity Index (MASI), the most commonly used outcome measure for melasma.
Quality of life analysis | 3 months
  Analysis of the quality of life of Melasma patients during the study will be performed using the MELASQol Instrument. It is a useful tool in assessing quality of life in patients with melasma.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana R dos Anjos Mendonça, PhD, Principal Investigator — Vale do Sapucaí University
Locations (1):
- Vale do Sapucaí University, Pouso Alegre, Minas Gerais, Brazil